CLINICAL TRIAL: NCT04892381
Title: Assessment of Programmed Cell Death Protein 1 (PD-1) and Programmed Cell Death Ligand 1 (PD-L1) Tissue Expression Levels in Lichen Planus Patients: A Case-Control Study
Brief Title: Assessment of PD-1 and PD-L1Tissue Expression Levels in Lichen Planus Patients: A Case-Control Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Fahim, Dermatology Lecturer, Cairo University
Other Study IDs: 13111993
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Lichen Planus
Keywords: LP; PD-1; PD-L1
MeSH Terms: conditions — Lichen Planus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lichen Planus group: Assessment of Programmed Cell Death Protein 1 (PD-1) and Programmed Cell Death Ligand 1 (PD-L1) Tissue Expression Levels using ELISA in lesional and non lesional skin
  Interventions: Diagnostic Test: Skin Biopsy
- Control group: Assessment of Programmed Cell Death Protein 1 (PD-1) and Programmed Cell Death Ligand 1 (PD-L1) Tissue Expression Levels using ELISA
  Interventions: Diagnostic Test: Skin Biopsy

INTERVENTIONS:
Diagnostic Test: Skin Biopsy — * Skin biopsy will be taken under local anesthesia :
  * From each normal control; a 3 mm punch skin biopsy from a sun protected area will be taken and preserved in PBS and kept frozen at -80 degrees Celsius for ELISA study.
  * From each LP patient; two punch skin biopsies will be taken and preserved in PBS and kept frozen at -80 degrees Celsius for ELISA study:
    i. The first biopsy will be a 3 mm punch biopsy from the center of LP lesional skin of sun protected area ii. The second biopsy will be a 3 mm punch biopsy from non lesional skin at least 15 cm away from the edge of any existing LP lesion of sun protected area
  * The level of PD1 and PD-L1 will be detected using ELISA technique.
  * The lesional biopsy will be assessed by routine hematoxylin and eosin (H&E) to confirm the diagnosis of LP

SUMMARY:
Assessment of Programmed Cell Death Protein 1 (PD-1) and Programmed Cell Death Ligand 1 (PD-L1) Tissue Expression Levels in Lichen Planus Patients: A Case-Control Study

DETAILED DESCRIPTION:
This prospective Case Control study will be conducted at Kasr Al-Aini Dermatology Outpatient Clinics and will include 30 LP patients and 30 normal healthy controls which will be recruited and assessed for eligibility for inclusion according to the above criteria.

All participants (patients & controls) will be subjected to the following:

* Written informed consent.
* Detailed history including onset, course, duration of the disease and history of drug intake within 1 month before the eruption.
* Clinical assessment of the Severity by using LP Severity Index (LPSI) (Kaur et al., 2020).
* Skin biopsy will be taken under local anesthesia :
* From each normal control; a 3 mm punch skin biopsy from a sun protected area will be taken and preserved in PBS and kept frozen at -80 degrees Celsius for ELISA study.
* From each LP patient; two punch skin biopsies will be taken and preserved in PBS and kept frozen at -80 degrees Celsius for ELISA study:

  i. The first biopsy will be a 3 mm punch biopsy from the center of LP lesional skin of sun protected area ii. The second biopsy will be a 3 mm punch biopsy from non lesional skin at least 15 cm away from the edge of any existing LP lesion of sun protected area
* The level of PD1 and PD-L1 will be detected using ELISA technique.
* The lesional biopsy will be assessed by routine hematoxylin and eosin (H&E) to confirm the diagnosis of LP
* Patients' serial numbers only will be used on data collection sheets and ELISA specimens' labels. Data will be entered on a computer with access limited to the researchers in order to ensure confidentiality of patients' information and lab results.

ELIGIBILITY:
Inclusion Criteria:

* Age group above 18 years old
* Patients of both genders
* Classic type of cutaneous LP.

Exclusion criteria:

* Topical treatment for LP 2 weeks before enrollment in the study or systemic treatment for LP 4 weeks before enrollment in the study and 3 years for systemic retenoids.
* Actinic LP , LP pigmentosus and Mucosal only LP
* Drug induced lichenoid eruption
* Conditions precluding taking skin biopsy : bleeding tendency , lidocaine allergy
* PD-1 associated-diseases e.g.: SLE, Cancers including melanoma and non-melanoma skin cancers, and Bullous Pemphigoid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 30 male and female Lichen Planus patients.
  * 30 male and female normal healthy Controls. Patients will be selected from Kasr Al-ainy, Dermatology Outpatient Clinic.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-18 (Estimated); Primary Completion 2022-04-18 (Estimated); Study Completion 2022-04-22 (Estimated)

PRIMARY OUTCOMES:
Measurement of the level of PD-1 and PD-L1 in the lesional and in non lesional skin in LP patients compared to normal controls | 12 months
  Programmed Cell Death Protein 1 (PD-1) and Programmed Cell Death Ligand 1 (PD-L1) Tissue Expression Levels in Lichen Planus Patients

CONTACTS AND LOCATIONS:
Overall Officials: Rana A Misaad, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elmasry MF, Mosaad RA, Azzam OA, Rashed LA, Fahim A. Assessment of PD-1 and PD-L1 tissue expression levels in lichen planus patients: a case-control study. Arch Dermatol Res. 2024 Mar 2;316(3):97. doi: 10.1007/s00403-024-02838-z. PMID 38430309